CLINICAL TRIAL: NCT03272399
Title: Targeted Alteration in Omega-3 and Omega-6 Fatty Acids for Post-traumatic Headache (Nutrition for PTH)
Brief Title: Nutrition for Post-Traumatic Headache
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Fort Belvoir Community Hospital (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency); University of North Carolina, Chapel Hill (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kimbra Kenney, Associate Professor, Neurology, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 416047
Record Dates: First submitted 2017-08-21; First posted 2017-09-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Post-Traumatic Headache Chronic Without Intractable Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H3-L6 (Experimental): High Omega-3, low Omega-6 diet
  Interventions: Other: Diet/nutrition intervention
- L3-H6 (Active Comparator): Control diet containing average US polyunsaturated fatty acid (PUFA) content with low omega-3 and high omega-6 content
  Interventions: Other: Diet/nutrition intervention

INTERVENTIONS:
Other: Diet/nutrition intervention — The intervention will be administered through food products rather than dietary supplements
  Other Names: High omega-3 versus high omega-6 dietary intervention

SUMMARY:
The purpose of this multi-site study is to evaluate the efficacy of a high omega-3/low omega-6 dietary intervention (the H3-L6 Diet) vs. a Control Diet in reducing headache pain and improving function in soldiers, veterans and military healthcare beneficiaries with post-traumatic headache (PTH). In addition, the study will examine the effects of the diet interventions on anti-nociceptive and pro-nociceptive lipid mediators derived from omega-3 and omega-6 fatty acids.

DETAILED DESCRIPTION:
Migraine-like PTH is an ideal patient population to test the effects of the H3-L6 intervention for several reasons. First, although PTH is considered a secondary headache syndrome, the fact that migraine-like PTH has a phenotype indistinguishable from primary migraine disorders and shares common pain-related comorbidities (e.g. anxiety, depression) suggests that shared biochemical mechanisms may underlie both conditions. Second, many PTH patients experience poor or incomplete therapeutic responses to available treatments, often while suffering from drug-related adverse effects. The prospect of improved headache outcomes with concurrent reduction in medication use (as seen in the Chronic Daily Headache Trial) may be particularly beneficial in PTH, since certain headache medications (e.g. opiates, muscle relaxants, sleep aids) have cognitive side effects, which may worsen residual cognitive impairment from Traumatic Brain Injury (TBI).

While PTH is an important cause of disability after TBI, problems with memory, executive function, depression, anxiety, irritability, fatigue, post-traumatic stress, and other neurobehavioral disorders are also common after TBI and contribute to disability. The H3-L6 (High Omega-3 Low Omega-6) intervention increased circulating concentrations of several key bioactive mediators which could hypothetically also have favorable effects on these TBI-associated non-headache impairments associated with TBI combat injuries. Omega-3 fatty acids have been widely studied in pre-clinical models and human TBI and demonstrate promising evidence of both neuroprotective and neurorestorative efficacy.

Potential mechanisms include antioxidant, anti-inflammatory, and pro-neurogenic effects. In our pilot study, the H3-L6 intervention significantly increased circulating levels of docosahexaenoic acid-eicosapentaenoic acid (DHA-EPA) , a potent stimulator of neurite growth and synaptogenesis in hippocampus and other central nervous system (CNS) tissues. Corresponding increases in the synaptamide biosynthesis in central nervous system tissues could hypothetically assist cognitive and functional neurorecovery associated with traumatic brain injury. Further, the reduction of proinflammatory metabolites of omega-6 fatty acids may provide additional benefits beyond what can be achieved through omega-3 supplementation alone.

Study Type: Interventional, Phase 2, double blind Study Design: Allocation: Randomized, parallel group Masking: Double Blind (Participant, Investigator, Outcomes Assessor) Primary Purpose: Treatment

Primary Outcome Measures:

Hypothesis and Objective: The investigators will obtain support for the following hypotheses through three specific aims:

Specific Aim 1: To compare the efficacy of the H3-L6 Diet to the Control Diet, in reducing headache pain and improving headache-related quality of life.

Hypothesis 1: Compared to the Control Diet, the H3-L6 Diet will produce significant improvement in:

(1a) the Headache Impact Test-a headache-specific quality of life measure-Primary Clinical Outcome);

(1b) mean total Headache Hours per day; and

(1c) mean Severe Headache Hours per day.

Secondary Outcomes Measures:

Specific Aim 2: To evaluate whether the H3-L6 Diet can increase circulating anti-nociceptive omega-3 metabolites, and reduce pro-nociceptive omega-6 metabolites, in patients with Posttraumatic Headaches.

Hypothesis 2: Compared to the Control Diet, the H3-L6 Diet will produce significant increases in anti-nociceptive omega-3 metabolites including 17-hydroxy DHA (Primary Biochemical Aim), and reductions in pro-nociceptive omega-6 metabolites.

Other Outcomes Measures Specific Aim 3: To explore the potential of the H3-L6 intervention for improving non-headache TBI outcomes.

Hypothesis 3: Compared to the Control Diet, the H3-L6 Diet will produce significant improvement in:

(3a) non-headache pain; (3b) depression/anxiety; (3c) symptoms of post-traumatic stress disorder; (3d) cognitive function; (3e) sleep quality; and (3f) will significantly reduce the use of acute pain medications. Enrollment: Up to 300 total participants enrolled among the 3 military sites for 120 12-week diet completers

ELIGIBILITY:
Inclusion Criteria:

* In order to be included in the study, you must be a person of either gender who is at least 18 years of age, meets criteria of having had a traumatic brain injury, a physiological disruption of brain function, as manifested by at least one of the following:

  1. . Any period of loss of consciousness
  2. . Any loss of memory for events immediately before or after the accident
  3. . Any alteration of mental state at the time of the accident (e.g., feeling dazed, disoriented, and confused)
  4. . Focal neurologic deficits that may or may not be permanent.

     * Traumatically induced includes the head being struck, the head striking an object, or the brain undergoing an acceleration/deceleration movement (i.e. whiplash) without direct external trauma to the head.
* Meets Internation Classification of Headache Disorders-version III (ICHD-III) criteria for persistent post-traumatic headache which is defined as a headache of at least 3 months duration caused by a traumatic injury to the head.
* Meets ICHD-III criteria for episodic/chronic migraine, with or without aura (excepting exclusion for organic disease):

  1. . Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
  2. . Headache has at least 2 of the following characteristics:

     1. unilateral location
     2. pulsating quality
     3. moderate or severe pain intensity
     4. aggravation by or causing avoidance of routine physical activity (eg, walking or climbing stairs)
  3. . During headache at least 1 of the following:

     1. nausea and/or vomiting
     2. photophobia and phonophobia
* A potential candidate for this study must be under the care of a physician for headaches and have an incomplete response to standard headache treatments.
* Must have headache frequency of more than 8 days per month.
* Must have a headache history of more than 6 months
* Must be able to attend or remotely participate (by video conference or telephone) in seven dietitian counseling sessions, and adhere to diet supplied to study participants.
* Must be a Department of Defense (DoD) healthcare beneficiary and eligible to receive care at Walter Reed National Military Medical Center (WRNMMC), Fort Belvoir Community Hospital (FBCH) or Womack Army Medical Center (WAMC).

Exclusion Criteria:

* A person cannot be in this study if they have a history of specific food allergies, especially to fish, dairy or gluten.

Also exclusionary are:

* Pregnancy or anticipated pregnancy
* Aversion to eating fish
* History of organic brain disorder other than TBI (vasculitis, encephalitis, meningitis, brain tumor)
* Major medical illness such as malignancy, diabetes, autoimmune or immune deficiency disorders, history of stroke or myocardial infarction
* Anticipated deployment or move to alternate location in the next 16 weeks
* Inability to read and communicate in English
* Regular use of fatty acid containing supplements
* Active or recent (2 years) history of treatment for substance abuse
* Cognitive impairment that prevents understanding of the protocol and completion of study procedures including compliance with the diet, blood draws and maintaining a daily headache diary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Clinical Outcome: To compare the efficacy of the high omega-3/low omega-6 (H3-L6) diet to the low omega-3/high omega-6 (L3-H6) diet in reducing headache pain and improving headache-related quality of life. | The HIT-6 is administered at study visits at week 0 (enrollment), 4, 10, 12, 14, 16
  Up to 300 participants complete the Headache Impact Test (HIT-6)-a headache-specific quality of life measure 6 times while enrolled in the study. The primary outcome measure is the change in the HIT-6 scores at baseline and at the end of the diet intervention.
Primary Biochemical Outcome: To evaluate the effects of the H3-L6 and L3-H6 Diet on circulating fatty acids and bioactive metabolites. | Fasting blood draws at study visits at weeks 4, 10, 16
  All study participants will have blood drawn 3 times during the 16-week study for analysis of circulating fatty acids and their bioactive metabolites. The following fatty acids will be measured in each blood sample (ng or pg per mL): 17-hydroxy-DHA (docosahexaenoic acid), 18-Hydroxy-EPA (eicosapentaenoic acid), 9-HODE (hydroxyl-octadecadienoic acid), 13-ODE (octadecadienoic acid), 5-HETE (hydroxyl-eicosatetraenoic acid), 8-HETE, 9-HETE, 11-HETE. Changes in 17-hydroxy-DHA and related fatty acids levels between blood draws at baseline and at the end of the 12-week diet intervention will be compared with changes in headache frequency and severity at the same time points.

SECONDARY OUTCOMES:
To compare the efficacy of the high omega-3/low omega-6 (H3-L6) diet to the low omega-3/high omega-6 (L3-H6) diet in reducing headache pain. | Daily on-line diary entry during the 16-week study
  Up to 300 participants complete a headache diary daily while enrolled in the 16-week study. Participants record the total number of headache hours per day. The outcome measure is the change in the mean daily headache hours at baseline and at the end of the diet intervention between the H3-L6 and L3-H6 diet intervention groups.
To explore the potential of the H3-L6 intervention for improving non-headache pain outcomes. | Study visits at week 0 and 16
  Compared to the Control Diet, the H3-L6 Diet may produce significant improvement in non-headache pain. A survey of pain, the Total Body Pain Scale, will be administered at baseline and at the end of the 12-week diet intervention. The outcome measure is a reduction in non-headache pain as measured by the survey at baseline and at the end of the diet intervention.
To explore the potential of the H3-L6 intervention for decreasing acute pain medication usage | Daily on-line diary entry during the 16-week study
  Compared to the Control Diet, the H3-L6 Diet may produce significant improvement in: Use of acute pain medications. Participants will daily record all pain medications used in that 24-hour period. The outcome measure is the change in the acute pain medications sued at baseline and at the end of the diet intervention between the H3-L6 and L3-H6 diet intervention groups.
To explore the potential of the H3-L6 intervention for improving sleep quality | the PSQI is administered at weeks 4 and 16 of the study
  Compared to the Control Diet, the H3-L6 Diet may produce significant improvement in sleep quality. A sleep quality survey, the PSQI, will be administered at baseline at and the end of the 12-week diet intervention. The outcome measure is the change in the PSQI score at baseline and at the end of the diet intervention between the H3-L6 and L3-H6 diet intervention groups.
To explore the potential of the H3-L6 intervention for improving psychological distress (depression/anxiety) | Study visits at week 0 and 16
  The PROMIS-29, a survey of psychological distress (depression/anxiety), will be administered at baseline and at the end of the 12-week diet intervention. The outcome measure is a reduction in depression and/or anxiety as measured by the PROMIS-29 at baseline and at the end of the diet intervention.
To explore the potential of the H3-L6 intervention for improving symptoms of post-traumatic stress disorder (PTSD) | The PCL-C is administered at study visits at weeks 4 &16
  Compared to the Control Diet, the H3-L6 Diet may produce significant improvement in symptoms of post-traumatic stress disorder (PTSD). The PCL-C, a survey of post-traumatic stress symptoms, will be administered at baseline and at the end of the 12-week diet intervention. The outcome measure is the reduction in the PCL-C score at baseline and at the end of the diet intervention between the H3-L6 and L3-H6 diet intervention groups.
To explore the potential of the H3-L6 intervention for improving post-concussive symptoms. | NSI and GOS-E are administered at weeks 4 and 16.
  Compared to the Control Diet, the H3-L6 Diet may produce significant improvement in post-concussive symptoms. The Neurobehavioral Symptom Inventory (NSI) and the Glasgow Outcome Score-Extended (GOS-E) will be administered at baseline and at the end of the 12-week diet intervention. The outcome measure is a change in the NSI and GOS-E score at baseline and at the end of the diet intervention between the H3-L6 and L3-H6 diet intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kimbra Kenney, MD, Principal Investigator — Uniformed Services University of the Health Sciences; Chris Ramsden, MD, Study Director — National Institutes of Health (NIH); John Mann, MD, Study Director — UNC
Locations (3):
- United States (3):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army Medical Center (WAMC), Fort Bragg, North Carolina
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Study data to be uploaded into Federation Interagency Traumatic Brain Injury Repository (FITBIR) and made accessible after study is completed
Supporting Information: Study Protocol, CSR
Time Frame: After study is uploaded into FITBIR
Access Criteria: Through FITBIR

REFERENCES:
- [Background] Ramsden CE, Faurot KR, Zamora D, Suchindran CM, MacIntosh BA, Gaylord S, Ringel A, Hibbeln JR, Feldstein AE, Mori TA, Barden A, Lynch C, Coble R, Mas E, Palsson O, Barrow DA, Mann DJ. Targeted alteration of dietary n-3 and n-6 fatty acids for the treatment of chronic headaches: a randomized trial. Pain. 2013 Nov;154(11):2441-2451. doi: 10.1016/j.pain.2013.07.028. Epub 2013 Jul 22. PMID 23886520
- [Background] Ramsden CE, Faurot KR, Zamora D, Palsson OS, MacIntosh BA, Gaylord S, Taha AY, Rapoport SI, Hibbeln JR, Davis JM, Mann JD. Targeted alterations in dietary n-3 and n-6 fatty acids improve life functioning and reduce psychological distress among patients with chronic headache: a secondary analysis of a randomized trial. Pain. 2015 Apr;156(4):587-596. doi: 10.1097/01.j.pain.0000460348.84965.47. PMID 25790451
- [Derived] Faurot KR, Cole WR, MacIntosh BA, Dunlap M, Moore CB, Roberson B, Guerra M, Domenichiello AF, Palsson O, Rivera W, Nothwehr A, Arrieux J, Russell K, Jones C, Werner JK, Clark R, Diaz-Arrastia R, Suchindran C, Mann JD, Ramsden CE, Kenney K. Targeted dietary interventions to reduce pain in persistent post-traumatic headache among service members: Protocol for a randomized, controlled parallel-group trial. Contemp Clin Trials. 2022 Aug;119:106851. doi: 10.1016/j.cct.2022.106851. Epub 2022 Jul 13. PMID 35842107
- See also: Medline Plus related topic: Traumatic Brain Injury — http://www.medlineplus.gov/traumaticbraininjury.html
- See also: Medline Plus related topic: Post-traumatic headache — http://www.medlineplus.gov/headache.html
- See also: Medline Plus related topic: Migraine — http://www.medlineplus.gov/migraine.html